

# DOCUMENTO DE HOJA DE INFORMACIÓN AL PACIENTE Y CONSENTIMIENTO INFORMADO PARA INVESTIGACIÓN CLÍNICA QUE NO IMPLIQUE MUESTRAS BIOLÓGICAS

v.1\_2024

**TÍTULO DEL ESTUDIO:** EFICACIA ANALGESICA DEL BLOQUEO SERRATO INTERCOSTAL VERSUS INFILTRACION DE PUERTOS EN COLECISTECTOMIA LAPAROSCOPICA: ENSAYO CLÍNICO ALEATORIZADO

INVESTIGADOR PRINCIPAL: Mº Teresa Fernández Martin

SERVICIO / UNIDAD/ CENTRO DE SALUD: Anestesiologia HURH

GERENCIA: HOSPITAL UNIVERSITARIO RIO HORTEGA

TELÉFONO DE CONTACTO: 637571685 EMAIL:

tfernandez@saludcastillayleon.es

NOMBRE DE LA LÍNEA DE TRABAJO:

VERSIÓN DE DOCUMENTO: (Número de versión, fecha): V3. 26/05/25

### **HOJA DE INFORMACIÓN AL PACIENTE**

Nos dirigimos a usted para informarle sobre un estudio de investigación en el que se le invita a participar. El estudio ha sido aprobado por el Comité de Ética de la Investigación con medicamentos de las Áreas de Salud de Valladolid.

Nuestra intención es que usted reciba la información correcta y suficiente para que pueda decidir si acepta o no participar en este estudio.

Sea cual sea su decisión, el equipo investigador quiere agradecer su tiempo y atención.



#### 1) ¿Cuál es el objetivo del estudio?

El control adecuado del dolor en pacientes intervenidos de colecistectomía laparoscópica continúa centrando la atención de los anestesiólogos, debido a que, a pesar de ser una técnica poco invasiva, hemos observado que en ocasiones es bastante dolorosa.

Dentro de una estrategia multimodal, donde se administran de manera conjunta fármacos analgésicos por diferentes vías de administración (técnicas de anestesia regional, intravenoso...) y de diferentes familias, el objetivo del estudio se basa en comparar la eficacia de las técnicas anestésicas aplicadas en la cirugía laparoscópica de vesícula en nuestra práctica diaria, que consisten en Infiltración de puertos de inserción de trocares laparoscópicos previa a su inserción o en la realización del bloqueo serrato-intercostal tras la inducción anestésica.

En pacientes sometidos a colecistectomía laparoscópica se va a realizar una evaluación en cuanto a calidad de recuperación postoperatoria, control del dolor, ausencia de efectos adversos y facilidad de realización.

El objetivo principal del estudio es comprobar la eficacia de las técnicas aplicadas y si alguna de ellas es superior o no a la otra. Por si ello pudiera redundar en una modificación del tratamiento analgésico.

#### 2) ¿En qué consiste mi participación en el estudio?

Los resultados de estos estudios ayudarán probablemente a tratar de manera más precisa a los pacientes con una enfermedad como la suya. Se van a evaluar dos técnicas analgésicas utilizadas en cirugía laparoscópica de vesícula para evaluar si alguna de ellas es superior a la otra, a fin de realizar en ese caso, una modificación de la práctica habitual, con el fin de mejorar su recuperación.

Usted como paciente no debe de realizar ninguna acción suplementaria a la que implica el proceso de la cirugía, puesto que se trata de evaluar la práctica habitual. Su participación se le va a solicitar para la utilización de los datos recogidos en la hoja de evaluación, a fin de realizar un análisis. No se utilizarán ninguno de sus datos



personales, tan solo aquellos que hemos explicado junto a sus datos demográficos (edad, sexo y enfermedades asociadas)

#### Describir:

- El estudio tendrá la duración hasta completar el número de pacientes necesario para llegar a una conclusión
- Solo serán necesarias las pruebas habituales para la cirugía, que incluyen el preoperatorio y la evaluación posterior del dolor y de la calidad de recuperación siguiendo los estándares del servicio de anestesia
- Datos de salud a los que se acceden (por ejemplo, Historia Clínica de Medora o Jimena), pruebas diagnósticas, etc.

#### 3) Algunas consideraciones sobre su participación:

Es importante que Vd., como participante en esta línea de trabajo, conozca diferentes aspectos de su participación:

- A) Su participación es totalmente voluntaria y puede decidir no participar. Si decide participar, puede cambiar su decisión y retirar el consentimiento (revocación) en cualquier momento, sin que por ello se altere la relación con su profesional sanitario ni se produzca perjuicio alguno en su atención sanitaria.
- B) Puede plantear todas las dudas que considere sobre su participación en este estudio, dirigiéndose al investigador principal del mismo.
- C) Es posible que los estudios realizados aporten información relevante para su salud o para la sociedad. Puede que no obtenga ningún beneficio para su salud por participar en este estudio.
- D) No percibirá ninguna compensación económica o de otro tipo por su participación en el estudio.

#### 4) Información básica sobre Protección de Datos



De acuerdo con lo establecido en el Reglamento (UE) 2016/679 del Parlamento Europeo y del Consejo, de 27 de abril de 2016, relativo a la protección de las personas físicas en lo que respecta al tratamiento de datos personales y a la libre circulación de estos datos (RGPD) y la Ley Orgánica 3/2018 de 5 de diciembre, de Protección de datos Personales y garantía de derechos digitales (LOPDPGDD) y cualquier otra norma de desarrollo se relaciona la información sobre el tratamiento de los datos personales incorporados al fichero del proyecto de Investigación.

| | INFORMACIÓN BÁSICA SOBRE PROTECCIÓN DE DATOS |
|---|---|
| Responsable | HOSPITAL UNIVERSITARIO RIO HORTEGA |
| Finalidad | Desarrollo del proyecto de Investigación |
| Legitimación | Art 6.1.a) RGPD. Consentimiento expreso |
| Destinatarios | Los datos podrán ser utilizados por el grupo del investigador principal en estudios futuros de investigación |
| | relacionados con la línea de trabajo arriba expuesta. Dichos datos podrán ser cedidos a otros investigadores |
| | designados por el Investigador Principal para trabajos relacionados con esta línea. En ambos casos, se requiere |
| | autorización previa del CEIm de las Áreas de Salud de Valladolid |
| Transferencia de datos | No están previstas transferencias internacionales de los datos sin anonimizar a terceros países u organizaciones |
| | internacionales |
| Derechos | Tiene derecho de acceso, rectificación, supresión, limitación y oposición al tratamiento, en los términos de los |
| | artículos 15 a 23 del RGPD. Puede ejercer todos estos derechos ante el responsable del tratamiento. Puede |
| | ejercer todos estos derechos ante el Delegado de Protección de Datos, a través de la dirección de correo: |
| | dpd@saludcastillayleon.es. Puede presentar una reclamación ante la Agencia Española de Protección de Datos. |
| | Más información en: www.agpd.es |
| Consulta información | https://www.saludcastillayleon.es/transparencia/es/proteccion-datos-personales |



#### CONSENTIMIENTO INFORMADO DEL PACIENTE POR ESCRITO

**Título del Estudio:** \_\_ EFICACIA ANALGESICA DEL BLOQUEO SERRATO INTERCOSTAL VERSUS INFILTRACION DE PUERTOS EN COLECISTECTOMIA LAPAROSCOPICA: ENSAYO CLÍNICO ALEATORIZADO

| Centro donde se realiza el estudio: HURH |
|---|
| Yo, |
| (Nombre y apellidos del paciente) |
| ☐ He leído la información que me ha sido entregada. |
| ☐ He recibido la hoja de información que me ha sido entregada. |
| ☐ He podido hacer preguntas sobre el estudio. |
| ☐ He recibido suficiente información sobre el estudio. |
| ☐ He hablado del estudio con |
| (Nombre y apellidos del investigador) |
| ☐ Comprendo que mi participación es voluntaria. |
| ☐ Comprendo que puedo retirarme del estudio: |
| 1 Cuando quiera. |
| 2 Sin tener que dar explicaciones. |
| <ol> <li>3 Sin que esto repercuta en mis cuidados médicos.</li> </ol> |
| Por la presente, otorgo mi consentimiento informado y libre para participar en esta investigación. |
| Accedo a que los profesionales del centro donde se realiza el estudio contacten conmigo en el futuro en caso de que se necesite obtener nuevos datos o actualizar la información asociada al estudio: |
| ☐SI☐NO (marcar con una X lo que proceda) |
| Accedo a que los profesionales del centro donde se realiza el estudio contacten conmigo |
| en caso de que los estudios realizados sobre mis datos aporten información relevante |
| para mi salud o la de mis familiares: |
| ☐SI☐ NO (marcar con una X lo que proceda) |



Recibiré una copia firmada y fechada de esta hoja de información y consentimiento informado.

| FIRMA DEL PACIENTE<br>NOMBRE Y APELLIDOS:<br>FECHA: | FIRMA DEL INVESTIGADOR NOMBRE Y APELLIDOS: FECHA: |
|---|---|
| | DEL CONSENTIMIENTO INFORMADO CON EL INVESTIGADOR PRINCIPAL) |
| Yoconsentimiento de participación | revoco e en el estudio. |
| FIRMA DEL PACIENTE: | |
| NOMBRE Y APELLIDOS: FECHA: | |



## CONSENTIMIENTO INFORMADO DEL REPRESENTANTE LEGAL DEL PACIENTE POR ESCRITO

**Título del Estudio:** \_\_ EFICACIA ANALGESICA DEL BLOQUEO SERRATO INTERCOSTAL VERSUS INFILTRACION DE PUERTOS EN COLECISTECTOMIA LAPAROSCOPICA: ENSAYO CLÍNICO ALEATORIZADO

| Centro donde se realiza el estudio:HURH |
|---|
| Yo, |
| como representante legal, del paciente |
| ☐ He leído la información que me ha sido entregada. |
| ☐ He recibido la hoja de información que me ha sido entregada. |
| ☐ He podido hacer preguntas sobre el estudio. |
| ☐ He recibido suficiente información sobre el estudio. |
| ☐ He hablado del estudio con |
| (Nombre y apellidos del investigador) |
| ☐ Comprendo que mi participación es voluntaria. |
| ☐ Comprendo que puedo retirarme del estudio: |
| 1 Cuando quiera. |
| 2 Sin tener que dar explicaciones. |
| 3 Sin que esto repercuta en mis cuidados médicos. |
| Por la presente, otorgo mi consentimiento informado y libre para que mi representado participe en esta investigación. |
| Accedo a que los profesionales del centro donde se realiza el estudio contacten conmigo en el futuro en caso de que se necesite obtener nuevos datos sobre mi representado: |
| □SI□NO (marcar con una X lo que proceda) |
| Accedo a que los profesionales del centro donde se realiza el estudio contacten conmigo en caso de que los estudios realizados sobre los datos aporten información relevante para su salud o la de sus familiares: |
| □SI□ NO (marcar con una X lo que proceda) |



Recibiré una copia firmada y fechada de esta hoja de información y consentimiento informado.

| FIRMA DEL REPRESENTANTE | FIRMA DEL INVESTIGADOR |
|-------------------------|------------------------|
| NOMBRE Y APELLIDOS: | NOMBRE Y APELLIDOS: |
| FECHA: | FECHA: |

### REVOCACIÓN DEL CONSENTIMIENTO INFORMADO (CONTACTAR CON EL INVESTIGADOR PRINCIPAL)

| Yo, |
|---|
| como representante legal del paciente |
| revoco el consentimiento de participación en el estudio arriba firmado. |
| FIRMA DEL REPRESENTANTE |
| NOMBRE Y APELLIDOS: |
| FECHA: |